CLINICAL TRIAL: NCT05875090
Title: Screening Trial for Glaucomatous Optic Discs in Portugal
Brief Title: Glaucoma Portugal Screening Trial
Acronym: Glaucoma PoST
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar Universitário Lisboa Norte (Other)
Collaborators: Unidade Local de Saúde do Alto Minho (Other); ACES Lisboa Norte (Unknown); Equipa Regional dos Programas de Rastreio da Região de Saúde de Lisboa e Vale do Tejo (Unknown); ACES Alto Minho (Unknown)
Responsible Party: Principal Investigator, Luis Abegao Pinto, Prof. Dr., Centro Hospitalar Universitário Lisboa Norte
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 38/23
Record Dates: First submitted 2023-04-13; First posted 2023-05-25 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Glaucoma
Keywords: Screening
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: Two models of population-based glaucoma screening will be tested. Lisbon center will conduct screening using an Artificial-Intelligence software based on optic disc centered retinographies. The Minho center will conduct screening based on OCT-based findings on the retinal nerve fibre layer thickness (RNFL)
Who Masked: Outcomes Assessor
Masking Description: Two physicians (unrelated to any recruiting center) will have access to pseudonymized data, masked to both screening and hospital decisions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-enhanced Retinography-based screening (Experimental): Screening in Lisbon arm will be done by an Artificial Intelligence (AI) software reading an optic disc entered retinography. Outcome of this analysis is referral vs non-referral based on a pre-established threshold.
  IOP 24mmHg or higher will be also be referred, regardless of optics disc analysis
  Interventions: Diagnostic Test: Glaucoma Screening
- OCT-based screening (Active Comparator): Screening in the Minho arm will be done based on optic coherence Tomography (OCT) retinal nerve fibre layer thickness (RNFL). Existence of a single sector outside normal limits (>95%) will be considered referrable.
  IOP 24mmHg or higher will be also be referred, regardless of optics disc analysis
  Interventions: Diagnostic Test: Glaucoma Screening

INTERVENTIONS:
Diagnostic Test: Glaucoma Screening — Non-invasive diagnostic techniques will screen subjects in primary care setting for the existence of Glaucoma and categorised them in a binary system: referrable vs non-referrable to a Hospital-based Glaucoma Clinic

SUMMARY:
Two primary care-based screening systems will be used to identify subjects with referrable glaucoma to hospital care.

Subjects between 55 to 65 years old living in two primary care areas (urban area in Lisbon ; countryside setting in Minho) will be invited to a one-time assessment of optic disc and intraocular pressure (IOP).

Criteria for referral will differ between centers, with one arm (Lisbon) using an artificial intelligence (AI) reading software of the optic disc picture, the other (Minho) will base their referral based on optical coherence tomography (OCT) retinal nerve fibre layer abnormality.

A masked reading center will be established to set the ground truth for diagnosis.

This pilot screening trial will explore the level of agreement between both systems as well as their cost effectiveness and identify diagnostic composite scores that could maximize the screening process. Secondary analyses will include the identification of population characteristics that increase effectivity of screening process as well as determining the population less likely to adhere to screening programmes.

DETAILED DESCRIPTION:
Glaucoma diagnosis is currently based on opportunistic case finding, which makes the case for up to 50% of patients remaining undiagnosed. Diagnostic technology has been deemed efficient in diagnosing, but cost and (hospital) location acts as a barrier for effective screening for this asymptomatic disease with a low population-based prevalence

Portuguese National Strategy for Visual Health, published in 2018 asks for a pilot study aimed at a one-time intervention at the primary care setting at the age of 60 years to do both an optic disc analysis and an intraocular pressure (IOP) measurement as a screening system for glaucoma

Two Portuguese centers have applied for this pilot. An urban-based center (Lisbon) and a countryside center (Minho) will conduct an invitation-based screening for those registered in their global primary care area. Age range was increased to 55 to 65 to capture a spectrum of data, enabling to later refine the target population.

Screening Intervention will be the same in both centers. Both will assess reasons for undergoing or rejecting screening and demographic and ophthalmological-related parameters, including glaucoma family history and a known personal glaucoma diagnosis. IOP will be non-invasively checked by rebound tonometry and optic disc retinographies will be performed on both centers. The Minho arm will additionally perform an optical coherence tomography (OCT) on all subjects.

Decision to refer will be made on one (or both) two findings:

1. IOP of 24mmHg or higher
2. referrable glaucoma

The Lisbon arm will use an Artificial intelligence (AI) system to rank the retinography findings into a binary referrable vs non-referrable system, based on a pre-defined threshold (0.73).

The Minho arm will base their referral on the existence of optical coherence tomography (OCT) retinal nerve fibre layer abnormality (defined as one sector thickness being outside normal limits)

Subjects flagged as referrable will be sent to the hospital Glaucoma Clinic, where functional and structural examinations will be performed and a standard of care clinical decision will be made by the glaucoma expert.

A reading center, with two masked experts, will be established to determine an unbiased ground truth for the comparison analysis. Reading center will conduct analysis on 3 tier level:

First round will include masked fundus pictures of all recruited subjects from both centers (both positive and negative referrals).

Second Round will include all subjects from Minho arm, who will have both fundus picture and OCT data.

Third round will include data analysis from all positive referrals from both arms, which includes all clinical data from the CRF plus all hospital exams (excluding clinical impression).

Outcomes of the reading center will be twofold:

1. "Glaucoma diagnosis label"

1. "normal"
2. "glaucoma suspect"
3. "definite glaucoma" (which implies a glaucomatous visual field) 2) Score (0-100) of likeliness of definitive glaucoma Disagreements on any category will be solved by a third masked referee (in the case of the scoring system, a difference larger than 10% would be considered a disagreement)

ELIGIBILITY:
Inclusion Criteria:

* subjects age between 55 to 65 years old registered in the primary care area of either ACES Lisbon Norte (Lisbon arm) or in the area of ACES Alto Minho (Minho arm)
* willingness to sign an informed consent for the screening process

Exclusion Criteria:

- none

Poor quality in screening image will be included in the intention to treat analysis, but excluded from the diagnostic comparator outcome.

Patients with a known glaucoma diagnosis will not be excluded from the screening

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic agreement between referring decision and reading center decision | Duration of the study (8 months)
  Level of agreement will be done between referring decision and the ground truth as assessed by the reading center (normal, glaucoma suspect; definitive glaucoma). All subjects from both centers (referred and non-referred) will be reviewed.
  For a primary outcome analysis, the middle category (glaucoma suspect) will be pooled together with the normal diagnosis

SECONDARY OUTCOMES:
Comparison between level of agreement (with ground truth) from both screening models | Duration of the study (8 months)
  Analysis on the differences in agreement between the AI-based referral and the OCT RNFL based referral in terms of the three possible outcomes by the reading center (normal; glaucoma suspect and definite glaucoma).
Level of performance of agreement by number of diagnostic testing | Duration of the study (8 months)
  Reading center will conduct analysis on 3 tier level. First round will include masked fundus pictures of all recruited subjects from both centers (both positive and negative referrals). Second Round will include all subjects from Minho arm, who will have both fundus picture and OCT data. Final round will include data analysis from all positive referrals from both arms, which includes all clinical data from the CRF plus all hospital exams (excluding clinical impression).
Cost effective analysis of both screening models | Duration of the study (8 months)
  Cost effective analysis will be performed on each arm comparing direct screening costs, stage of visual impairment of patients detected through screening and the opportunity saving by the screening compared to a standard case-finding scenario (literature reference).
Subjects parameters associated with positive screening | Duration of the study (8 months)
  Analysis will be performed to explore a priori subjects characteristics that could be associated with a positive screening results (such as age, ethnic background, family history). Statistical models will be made to identify target population more likely to benefit from screening
Parameters associated with accepting screening system by the patients | Duration of the study (8 months)
  Analysis will be done on all contacted patients (including the ones who did not accept to undergo screening) to identify which are the populations less likely to enter a screening circuit
Level of agreement (in %) between AI-risk score and human-based assessment of disease severity | Duration of the study (8 months)
  Reading center risk score of disease severity (ranked from 0 to 100) will be compared to the AI-based disease score. This will be done separately in each of the 3 categories (normal; glaucoma suspect; glaucoma). Analysis of this score would help refine clinical risk (high risk vs low risk patients) of each category. Exploratory analysis will be made to determine the added value of including this risk score in refining AI-based referral

CONTACTS AND LOCATIONS:
Overall Officials: Luis Abegão Pinto, MD, PhD, Study Chair — Centro Hospitalar Universitário Lisboa Norte; Sérgio Azevedo, MD, Study Chair — Unidade Local Saude Alto Minho
Locations (3):
- Portugal (3):
  - Equipa Regional dos Programas de Rastreio da Região de Saúde de Lisboa e Vale do Tejo, Lisbon
  - Centro Hospitalar Lisbon Norte, Lisbon
  - Unidade Local Saude Alto Minho, Viana do Castelo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] US Preventive Services Task Force; Mangione CM, Barry MJ, Nicholson WK, Cabana M, Chelmow D, Coker TR, Davis EM, Donahue KE, Epling JW Jr, Jaen CR, Krist AH, Kubik M, Li L, Ogedegbe G, Pbert L, Ruiz JM, Simon MA, Stevermer J, Wong JB. Screening for Primary Open-Angle Glaucoma: US Preventive Services Task Force Recommendation Statement. JAMA. 2022 May 24;327(20):1992-1997. doi: 10.1001/jama.2022.7013. PMID 35608574
- [Background] Hemelings R, Elen B, Barbosa-Breda J, Lemmens S, Meire M, Pourjavan S, Vandewalle E, Van de Veire S, Blaschko MB, De Boever P, Stalmans I. Accurate prediction of glaucoma from colour fundus images with a convolutional neural network that relies on active and transfer learning. Acta Ophthalmol. 2020 Feb;98(1):e94-e100. doi: 10.1111/aos.14193. Epub 2019 Jul 25. PMID 31344328
- [Background] Sousa DC, Leal I, Nascimento N, Marques-Neves C, Tuulonen A, Abegao Pinto L. Use of Ocular Hypotensive Medications in Portugal: PEM Study: A Cross-sectional Nationwide Analysis. J Glaucoma. 2017 Jun;26(6):571-576. doi: 10.1097/IJG.0000000000000668. PMID 28368997